CLINICAL TRIAL: NCT04013451
Title: Kindness as an Intervention for Student Social Interaction Anxiety, Resilience, Affect, and Mood
Brief Title: The Kiss of Kindness Study II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Jennifer Irwin, Full-time Professor, Faculty of Health Sciences, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114103
Record Dates: First submitted 2019-06-28; First posted 2019-07-09 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Anxiety; Stress; Mood; Affect
Keywords: kindness; social interaction anxiety; mood; affect; resilience; undergraduate students; graduate students
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants allocated to the intervention group will participate in the intervention (acts of kindness).
  Interventions: Behavioral: Acts of kindness
- Control Group (No Intervention): Participants allocated to the control group will not participate in the intervention and will act as the comparison condition.

INTERVENTIONS:
Behavioral: Acts of kindness — Both intervention and control groups will receive an email with access to a relaxation and stress management booklet from Western University's (UWO) Wellness Education Centre (http://studentexperience.uwo.ca/docs/RelaxationAndStressManagement.pdf). In addition, the intervention group will be asked to (1) complete and log/submit a minimum of three deliberate acts of kindness per day for one month, and (2) join the study-dedicated online site to connect with, support, and share experiences and ideas with each other around acts of kindness.
  Arms: Intervention Group

SUMMARY:
The objective of this study is to assess the impact of engaging in deliberate acts of kindness on resilience (primary outcome); social interaction anxiety and affect (secondary outcomes); and mood (exploratory outcome) of undergraduate and graduate students at Western University (UWO). Recruitment of 200 participants consisting of 150 full-time undergraduate and 50 graduate students, randomized to either the intervention (n=100) or control group (n=100) will be achieved via a mass email to all full-time students at UWO. Both intervention and control groups will receive an email with access to a relaxation and stress management booklet from UWO's Wellness Education Centre (http://studentexperience.uwo.ca/docs/RelaxationAndStressManagement.pdf). In addition, the intervention group will be asked to (1) complete and log/submit a minimum of three deliberate acts of kindness per day for one month, and (2) join the study-dedicated online site to connect with, support, and share experiences and ideas with each other around acts of kindness. Individuals in the intervention group will also receive a list of deliberate acts of kindness ideas, for reference. Baseline, immediate post intervention, and three-months post intervention data will be collected using previously validated questionnaires associated with each outcome of interest, and posted to Qualtrics, an online survey tool. Additionally, immediately following the intervention and 3 months post intervention all participants will complete an open-ended question asking them to describe their overall experience being involved in the study. Quantitative and qualitative data analysis will occur upon the completion of the study.

DETAILED DESCRIPTION:
Poor mental health is a significant public health concern that disproportionally affects university students, compared to their community counterparts, and stress is a main culprit. Although privileged in terms of attending higher education, the stress-related inequity experienced among university students stems from "academic load, constant pressure to succeed, competition with peers, financial burdens, and peer, teacher or parental pressure". These stressors can trigger or exacerbate anxiety levels, which are on the rise among students. The most recent National College Health Assessment Survey, which included Canadian postsecondary institutions, showed a marked increase in student anxiety between 2013 to 2016. Although less studied than undergraduates, graduate students' mental health also is worrisome with over 60% feeling exhausted, overwhelmed, hopeless, and/or depressed nearly all of the time. It is imperative that evidence-informed approaches to enhance resilience and reduce the negative mental health experiences of undergraduate and graduate students be implemented and evaluated. Although improving resilience and overall mental health is a growing focus across campuses, current programming is clearly unable to address the concern in its entirety, and additional interventions are required.

An emerging and promising approach to promoting positive mental health and resilience among secondary students is performing acts of kindness. Arguably, performing acts of kindness improves mental health through the strengthening of psychological resilience. Resilience, as an outcome, is predicated on six underlying dimensions: health, collaboration, purpose, composure, reasoning, and tenacity. In terms of health and collaboration, a small classroom-based kindness pilot entailing logging acts of kindness by undergraduate students at Western University (UWO), found improvements in individual levels of wellbeing (i.e. confidence and decreased stress), perceptions of positive classroom culture, and classroom cohesion. Performing acts of kindness is correlated with happiness which results in a positive sense of purpose, increased composure, and improved reasoning and resilience. Moreover, the physiological effects are well-known as functional magnetic resonance images (fMRIs) show activation in the reward centres of the brain when subjects are engaged in acts of kindness. Despite the strong theoretical foundation that links acts of kindness with resilience, this area of research has yet to be sufficiently explored. To that end, the objective of this study is to assess the impact of engaging in deliberate acts of kindness on resilience (primary outcome); social interaction anxiety and affect (secondary outcomes); and mood (exploratory outcome) of undergraduate and graduate students at UWO.

Methods

Study Design

A longitudinal repeated-measures, mixed methods randomized control trial grounded in an interpretive description paradigm will be used. Interpretive description is an inductive analysis approach that creates ways of understanding phenomena yielding application-based implications for practice. Recruitment of 200 participants consisting of 150 full-time undergraduate and 50 graduate students, randomized to either the intervention (n=100) or control group (n=100) will be achieved via a mass email to all full-time students at UWO once ethical approval is obtained and the trial is registered. This sample size was selected considering two criteria: 1) based on our previous work in the area the sample size is feasible; and 2) from a power analysis using resilience as the primary outcome, a sample of 100 per group is sufficient to detect significant differences between groups (p < 0.05). Participants will be eligible if they are: (a) full-time undergraduate or graduate students at UWO and/or the affiliate schools (Kings, Brescia, Huron) and (b) English-speaking. Both intervention and control group participants will receive an email with access to a relaxation and stress management booklet from UWO's Wellness Education Centre. In addition, the intervention group will be asked to (1) complete and log/submit a minimum of three deliberate acts of kindness per day for one month, and (2) join the study-dedicated online site to connect with, support, and share experiences and ideas with each other around acts of kindness. Deliberate acts of kindness will be defined for participants as purposeful acts benefitting others that the others would presumably like.

Data Collection/Metrics

Baseline, immediate post intervention, and three-months post intervention data will be collected using Qualtrics, an online survey tool. Baseline will consist of basic demographic information, and four previously validated scales: (1) Brief Resilience Scale (BRS); (2) Social Interaction Anxiety Scale-Straightforward (SIAS-S); (3) International Positive and Negative Affect Schedule-Short Form (I-PANAS-SF); and (4) Brief Mood Introspection Scale (BMIS). The assessments will take 15-minutes to complete. After the completion of the baseline assessment participants will be randomized using stratification by degree level (i.e., undergraduate or graduate). Immediately following the intervention and 3 months post intervention all participants will complete the same assessments administered at baseline (minus demographics) with the addition of an open-ended question asking participants to describe their overall experience being involved in the study.

Data analysis

Data analysis will occur upon the completion of the study and quantitative data analysis will initially involve computing measures of central tendency and dispersion as well as the computation of the validated scales. Next, general linear models will be used to examine both differences between groups and overtime. For the qualitative data, inductive content analysis using interpretive description will be conducted independently, and simultaneously by two researchers who will subsequently meet, upon the completion of analysis, to determine agreement in emerging findings. Statistical Package for Social Sciences (SPSS) will be used for quantitative analysis and QSR International NVivo software will be used to code and categorize qualitative data. Knowledge Translation will involve both traditional mechanisms (publications/conferences) and engagement with social media (infographics, youtube videos).

ELIGIBILITY:
Inclusion Criteria:

* full-time undergraduate or graduate students at Western University (UWO) and/or the affiliate schools (Kings, Brescia, Huron)
* English-speaking

Exclusion Criteria:

* non-English-speaking (i.e. unable to understand and complete surveys/questionnaires)
* part-time students

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Resilience (Brief Resilience Scale) | Change from baseline resilience at immediate post-intervention and 3-month post-intervention
  The Brief Resilience Scale (BRS) includes 6-items; items 1, 3, and 5 are positively worded and items 2, 4, and 6 are negatively worded. Participants will be asked the extent to which they agree or disagree with the statements using a 5-point scale; 1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, and 5 = strongly agree. The BRS is scored by reverse coding items 2, 4, and 6, such that 5 = strongly disagree, 4 = disagree, 3 = neutral, 2 = agree, and 1 = strongly agree. The mean of the six items is then determined to score the scale.

SECONDARY OUTCOMES:
Social interaction anxiety (Social Interaction Anxiety Scale-Straightforward) | Change from baseline social interaction anxiety at immediate post-intervention and 3-month post-intervention
  The Social Interaction Anxiety Scale-Straightforward (SIAS-S) includes 20 items assessing cognitive, affective and behavioural aspects of social interaction anxiety using a five-point scale; 0 = not at all, 1 = slightly, 2 = moderately, 3 = very and 4 = extremely. Participants will be asked to indicate the degree to which they feel the statement is characteristic or true to them. The SIAS-S uses reverse coding, such that items 5, 9 and 11 are reverse scored; however, they are not included in the total score. A total score of 28 or higher indicates probable social interaction anxiety.
Affect (International Positive and Negative Affect Schedule-Short Form) | Change from baseline affect at immediate post-intervention and 3-month post-intervention
  The International Positive and Negative Affect Schedule-Short Form (I-PANAS-SF) includes 20 items from the Positive and Negative Affect Schedule (10 items = positive affect; 10 items = negative affect) using a five-point scale; 1 = very slightly or not at all, 2 = a little, 3 = moderately, 4 = quite a bit and 5 = extremely. Participants will be asked to indicate the extent they have felt the adjective over the past week. The positive affect score is obtained by adding the scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17 and 19. The negative affect score is obtained by adding the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18 and 20.

OTHER OUTCOMES:
Mood (Brief Mood Introspection Scale) | Change from baseline mood at immediate post-intervention and 3-month post-intervention
  The Brief Mood Introspection Scale (BMIS) is a mood-adjective scale that includes 16-items selected from eight mood states: (a) happy (happy, lively), (b) loving (loving, caring), (c) calm (calm, content), (d) energetic (active, peppy), (e) fearful/anxious (jittery, nervous), (f) angry (grouchy, fed up), (g) tired (tired, drowsy), and (h) sad (gloomy, sad). Participants will be asked to indicate how well each adjective or phrase describes their present mood. To score the BMIS, the numerical values from 1 to 4 are assigned to the Likert scale; 1 = definitely do not feel, 2 = do not feel, 3 = slightly feel and 4 = definitely feel, for both the positive and negative mood adjectives. Reverse scoring is used in order to accurately depict the participant's mood. To reverse score the BMIS, the numerical values assigned previously are reversed, such that 4 = definitely do not feel and 1 = definitely feel.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Irwin, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be disseminated via publications and presentations.
Supporting Information: Study Protocol
Time Frame: The intervention will take place during the month of November 2019 and the trial protocol will be submitted for publication; manuscript preparation will occur starting April 2020.

REFERENCES:
- [Background] Patel V, Flisher AJ, Hetrick S, McGorry P. Mental health of young people: a global public-health challenge. Lancet. 2007 Apr 14;369(9569):1302-1313. doi: 10.1016/S0140-6736(07)60368-7. PMID 17434406
- [Background] Dachew BA, Azale Bisetegn T, Berhe Gebremariam R. Prevalence of mental distress and associated factors among undergraduate students of University of Gondar, Northwest Ethiopia: a cross-sectional institutional based study. PLoS One. 2015 Mar 20;10(3):e0119464. doi: 10.1371/journal.pone.0119464. eCollection 2015. PMID 25794278
- [Background] Adlaf EM, Gliksman L, Demers A, Newton-Taylor B. The prevalence of elevated psychological distress among Canadian undergraduates: findings from the 1998 Canadian Campus Survey. J Am Coll Health. 2001 Sep;50(2):67-72. doi: 10.1080/07448480109596009. PMID 11590985
- [Background] Association, American College Health, E. (2016). ACHA - National College Health Assessment II: Ontario Canada Reference Group Executive Summary Spring 2016. American College Health Association, 1-18.
- [Background] Evans TM, Bira L, Gastelum JB, Weiss LT, Vanderford NL. Evidence for a mental health crisis in graduate education. Nat Biotechnol. 2018 Mar 6;36(3):282-284. doi: 10.1038/nbt.4089. No abstract available. PMID 29509732
- [Background] Paviglianiti, N. C., & Irwin, J. D. (2017). Students ' Experiences of a Voluntary Random Acts of Kindness Health Promotion Project, 1(August), 1-23
- [Background] Lyubomirsky, S., & Della Porta, M. D. (2010). Boosting happiness, buttressing resilience. Handbook of adult resilience, 450-464.
- [Background] Rossouw, P. J., & Rossouw, J. G. (2016). The predictive 6-factor resilience scale: Neurobiological fundamentals and organizational application. International Journal of Neuropsychotherapy, 4(1), 31-45.
- [Background] Lyubomksky, S., Sheldon, K. M., & Schkade, D. (2005). Pursuing happiness: The architecture of sustainable change. Review of General Psychology, 9(2), 111-131. https://doi.org/10.1037/1089-2680.9.2.111
- [Background] Cutler J, Campbell-Meiklejohn D. A comparative fMRI meta-analysis of altruistic and strategic decisions to give. Neuroimage. 2019 Jan 1;184:227-241. doi: 10.1016/j.neuroimage.2018.09.009. Epub 2018 Sep 7. PMID 30195947
- [Background] Thorne, S., Kirkham, S. R., & O'Flynn-Magee, K. (2004). The analytic challenge in interpretive description. International journal of qualitative methods, 3(1), 1-11.
- [Background] The Unviersity of Western Ontario (N.D.). Relaxation and Stress Management. http://studentexperience.uwo.ca/docs /RelaxationAndStress Management.pdf
- [Background] Trew, J. L., & Alden, L. E. (2015). Kindness reduces avoidance goals in socially anxious individuals. Motivation and emotion, 39(6), 892-907.
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Mayer JD, Gaschke YN. The experience and meta-experience of mood. J Pers Soc Psychol. 1988 Jul;55(1):102-11. doi: 10.1037//0022-3514.55.1.102. PMID 3418484
- [Background] Patton, M. Q. (2002). Two decades of developments in qualitative inquiry: A personal, experiential perspective. Qualitative social work, 1(3), 261-283.